CLINICAL TRIAL: NCT00107016
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled, Multi-center Study Assessing the Value of Adding Everolimus to Letrozole as Preoperative Therapy of Primary Breast Cancer in Postmenopausal Women
Brief Title: Everolimus and Letrozole as Preoperative Therapy of Primary Breast Cancer in Post-menopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRAD001C2222
Record Dates: First submitted 2005-04-04; First posted 2005-04-05 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-02

CONDITIONS: Breast Neoplasm
Keywords: Breast Cancer; Cancer of the Breast; Neo-adjuvant; Primary breast cancer; postmenopausal; pre-operative
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Letrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- RAD001 + letrozole 2.5mg (Experimental)
  Interventions: Drug: RAD001, Letrozole 2.5mg
- Letrozole 2.5mg (Active Comparator)
  Interventions: Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: RAD001, Letrozole 2.5mg
  Arms: RAD001 + letrozole 2.5mg
Drug: Letrozole 2.5mg
  Arms: Letrozole 2.5mg

SUMMARY:
The purpose of this study is to examine the effect of the combination of everolimus and letrozole compared to placebo and letrozole as pre-surgical therapy in patients with newly diagnosed estrogen receptor positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed diagnosis of invasive breast cancer, previously untreated
* Patients must be postmenopausal
* Candidates for mastectomy or breast-conserving surgery
* Primary tumor of above 2 cm diameter, measured by imaging
* Clinical Stage M0
* WHO performance status ≤1
* Adequate bone marrow, liver, and renal function

Exclusion Criteria:

* Multicentric invasive tumors
* Bilateral or inflammatory breast cancer
* Receiving concomitant anti-cancer treatments such as chemotherapy
* Patients with an uncontrolled infection
* Patients with other concurrent severe and/or uncontrolled medical disease

Additional protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2005-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To assess the added efficacy obtained by combining RAD001 and letrozole as preoperative therapy for four months in hormone-receptor positive breast cancer in postmenopausal women

SECONDARY OUTCOMES:
To assess the four month treatment as being predictive of clinical tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- United States (10):
  - Highlands Oncology Group, Springdale, Arkansas
  - Breastlink Medical Group Inc., Long Beach, California
  - UCSF Breast Care Center, San Francisco, California
  - University of Miami, Miami, Florida
  - Loyola University Medical Center, Maywood, Illinois
  - Investigative Clinical Research of Indiana, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - UPMC / Magee Womens Hospital, Pittsburgh, Pennsylvania
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Wilrijk, Belgium
- Canada (2):
  - Novartis Investigative Site, Natasha
  - Novartis Investigative Site, Winnipeg
- France (5):
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Saint-Herblain
- Germany (8):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankurt Am Main
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Tübingen
- Italy (4):
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Naples
  - Novartis Investigative Site, Torino
- Russia (3):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Saint Petersburg
- Spain (6):
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Zaragoza
- United Kingdom (5):
  - Novartis Investigative Site, Chelmsford
  - Novartis Investigative Site, Edinburgh
  - Novartis Investigative Site, Epping
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Whittington

REFERENCES:
- [Derived] Baselga J, Semiglazov V, van Dam P, Manikhas A, Bellet M, Mayordomo J, Campone M, Kubista E, Greil R, Bianchi G, Steinseifer J, Molloy B, Tokaji E, Gardner H, Phillips P, Stumm M, Lane HA, Dixon JM, Jonat W, Rugo HS. Phase II randomized study of neoadjuvant everolimus plus letrozole compared with placebo plus letrozole in patients with estrogen receptor-positive breast cancer. J Clin Oncol. 2009 Jun 1;27(16):2630-7. doi: 10.1200/JCO.2008.18.8391. Epub 2009 Apr 20. PMID 19380449